CLINICAL TRIAL: NCT07122427
Title: Aging of the Vascular Wall
Acronym: VITAL
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN502025/CHUSTE
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Vascular Risk; Aging Disorder
Keywords: Cardiovascular diseases; Aging; Eendothelial dysfunction
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Youngs: Patients aged 18 to 30 requiring coronary artery bypass grafting (CABG).
  Interventions: Procedure: Graft collection
- Middle-aged: Patients aged 30 to 60 requiring coronary artery bypass grafting (CABG).
  Interventions: Procedure: Graft collection
- Elderly: Patients aged 60 and more requiring coronary artery bypass grafting (CABG).
  Interventions: Procedure: Graft collection

INTERVENTIONS:
Procedure: Graft collection — Sampling of superior venous and arterial grafts (internal mammary artery, great saphenous vein) after coronary artery bypass surgery.

SUMMARY:
Demographic aging is predicted to be one of the most significant social changes of the 21st century. Aging is a slow, multifactorial process that progressively impacts the integrity of cells, tissues, and organs. This decline in function increases the risk of numerous diseases, including cancer, neurodegenerative disorders, and cardiovascular diseases (CVD). CVD, the leading global cause of death, becomes more prevalent with age. Aging contributes to endothelial dysfunction, vessel stiffness, thickening, and impaired platelet function. These changes disrupt hemostatic processes and increase the risk of cardiovascular complications. Despite preventive strategies CVD remain a major public health challenge. Cellular aging, or senescence, affects all cell types, particularly endothelial cells and platelets. However, little research has compared the aging rates of different blood vessel types, such as arteries and veins. Given their distinct compositions and developmental origins, it is likely that their aging processes differ at molecular, cellular, and physiological levels.

ELIGIBILITY:
Inclusion Criteria:

* Major patients requiring coronary artery bypass grafting (CABG).

Exclusion Criteria:

* Hypertension, diabetes, systemic inflammatory disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring coronary artery bypass grafting (CABG).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of ageing | Day 1
  Detection of innovative biomarkers of ageing by microscope analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore CAMPISI, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France, France

IPD SHARING:
Plan to Share IPD: No